CLINICAL TRIAL: NCT06310018
Title: A Prospective, Single-Arm, Multicenter Study of Augmented Ultrasound-Facilitated, Catheter-Directed Low-Dose Fibrinolysis for Pulmonary Embolism (SONIC-PE)
Brief Title: Augmented Ultrasound-Facilitated, Catheter-Directed Fibrinolysis for PE
Acronym: SONIC-PE
Status: Suspended | Type: Observational
Why Stopped: Awaiting completion and reporting of related trial
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2023A070902
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism; Right Ventricular Dysfunction; Right Ventricular Failure
Keywords: pulmonary embolism; right ventricular failure; right ventricular dysfunction; catheter-directed therapy; fibrinolysis
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right; Heart Failure | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ultrasound-facilitated, catheter-directed lower-dose fibrinolysis: 10 patients with bilateral PE will be treated with ultrasound-facilitated, catheter-directed lower-dose fibrinolysis (total dose 8 mg tPA given as 2 mg/hour/catheter over 2 hours) followed by 50 patients (total dose 6 mg tPA given as 3 mg/hour/catheter given over 1 hour) with the EKOS+™ system
  Interventions: Device: Ultrasound-facilitated, catheter-directed lower-dose fibrinolysis; Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Device: Ultrasound-facilitated, catheter-directed lower-dose fibrinolysis — Ultrasound-facilitated, catheter-directed lower-dose fibrinolysis (treated with a total dose 8 mg tPA given as 2 mg/hour/catheter over 2 hours for first 10 patients followed by 50 patients treated with total dose 6 mg tPA given as 3 mg/hour/catheter given over 1 hour) with the EKOS+™ system
Drug: Tissue Plasminogen Activator — total dose 8 mg tPA given as 2 mg/hour/catheter over 2 hours for first 10 patients followed by 50 patients treated with total dose 6 mg tPA given as 3 mg/hour/catheter given over 1 hour

SUMMARY:
SONIC-PE is a multicenter, prospective, single-arm study of 10 patients with bilateral PE treated with ultrasound-facilitated, catheter-directed lower-dose fibrinolysis (total dose 8 mg tPA given as 2 mg/hour/catheter over 2 hours) followed by 50 patients (total dose 6 mg tPA given as 3 mg/hour/catheter given over 1 hour) with the EKOS+™ system to determine its impact on the change in RV-to-LV diameter, refined Modified Miller Score, and distal pulmonary vascular blood volume as well as to assess International Society on Thrombosis and Haemostasis (ISTH) major bleeding.

DETAILED DESCRIPTION:
Patients with intermediate-high risk pulmonary embolism (PE) comprise a population at increased risk for clinical deterioration despite initially stable hemodynamics. The pathophysiology of hemodynamic deterioration in intermediate-high risk PE includes an abrupt increase in pulmonary vascular resistance, due to proximal as well as distal pulmonary artery occlusion, pulmonary hypertension, right ventricular (RV) pressure overload, and, ultimately, RV failure. While full-dose systemic fibrinolysis for PE has demonstrated efficacy for prevention of early morbidity and mortality, its net clinical benefit is attenuated by the risk of major bleeding, in particular intracranial hemorrhage. Catheter-directed therapies have been demonstrated to facilitate RV recovery while reducing the risk of major bleeding through use of lower-dose fibrinolysis or avoiding it altogether. Specifically, lower-dose regimens for ultrasound-facilitated, catheter-directed fibrinolysis result in sustained recovery of echocardiographically-determined RV function, reduction in Modified Miller Score (large-vessel pulmonary angiographic obstruction), functional status, and quality of life over the year following ultrasound-facilitated, catheter-directed fibrinolysis.

Recently, an upgrade to the output of the ultrasonic core catheter of the EKOS™ Endovascular System (EKOS+™) has demonstrated the ability to enhance fibrinolysis within a lower fibrinolytic dose range in preliminary studies (Boston Scientific Corporation, Maple Grove, MN). Compared with current EkoSonic™ system, a 50% increase in ultrasound power (measured in watts) with EKOS+™ resulted in a 130% increase in in vitro clot lysis compared with conventional catheter-directed fibrinolysis using the same dose of fibrinolytic drug.

SONIC-PE is multicenter, prospective single-arm study of 10 patients with bilateral PE treated with ultrasound-facilitated, catheter-directed lower-dose fibrinolysis (total dose 8 mg tPA given as 2 mg/hour/catheter over 2 hours) followed by 50 patients (total dose 6 mg tPA given as 3 mg/hour/catheter given over 1 hour) with the EKOS+™ system to determine its impact on the change in RV-to-LV diameter, refined Modified Miller Score, and distal pulmonary vascular blood volume as well as assess International Society on Thrombosis and Haemostasis (ISTH) major bleeding. The study will have an adaptive design component with transition to 8 mg tPA/2 hours if there is an excess of bleeding or observed lack of efficacy, as determined by an Independent Study Safety Monitor.

ELIGIBILITY:
Inclusion Criteria:

1. patients at least 18 years of age,
2. symptomatic PE defined as symptoms for <14 days with normal systolic blood pressure (>90 mmHg), RV-to-LV diameter ratio ≥0.9 on initial chest CT, bilateral filling defects located in at least 1 main or proximal lobar pulmonary artery, and cardiac troponin greater than the upper limit of normal (cTnI, cTnT, hsTnI, or hsTnT), AND
3. in whom ultrasound-facilitated, catheter-directed lower-dose fibrinolysis has been selected for treatment on a clinical basis.

Exclusion Criteria:

1. stroke or transient ischemic attack, head trauma, other active intracranial or intraspinal disease (including malignancy) within 1 year
2. recent active bleeding from a major organ within 1 month
3. major surgery within 7 days of screening
4. contraindication to therapeutic anticoagulation
5. systolic blood pressure <90 mm Hg, systolic blood pressure drop by at least 40 mmHg over at least 15 minutes, shock, use of vasopressors, need for CPR, or need for ECMO
6. need for mechanical ventilation, including non-invasive positive pressure ventilation
7. hematocrit <30%, platelet count <100,000/μl
8. international normalized ratio >3
9. serum creatinine > 2 mg/dL
10. liver cirrhosis
11. known hypersensitivity to tPA, heparin, or any excipients
12. perceived high risk for fatal or catastrophic bleeding
13. prescription of dual antiplatelet therapy (DAPT) at time of screening
14. Patients treated with any other advanced therapy, such as surgical embolectomy, catheter-based mechanical embolectomy, or fibrinolytic therapy, within the prior 30 days
15. pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present for evaluation and treatment of PE and in whom the decision to proceed with the EKOS+™ ultrasound-facilitated, catheter-directed lower-dose fibrinolytic procedure will be screened for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in RV-to-LV diameter ratio as measured by chest CT from baseline to 48 ± 6 hours | 48 ± 6 hours
  Change in RV-to-LV ratio will be determined by a dedicated core imaging laboratory, blinded to clinical data and timing of the CT studies
Frequency of ISTH major bleeding at 72 hours | 72 hours
  Adjudicated independently using ISTH criteria

SECONDARY OUTCOMES:
Change in chest CT-measured blood volume in the distal pulmonary vasculature from baseline to 48 ± 6 hours | 48 ± 6 hours
  Baseline and 48 ± 6 hours CT scans will be analyzed offline using 3D volumetric analysis
Change in refined Modified Miller Score as measured by chest CT from baseline to 48 ± 6 hours as measured by chest CT from baseline to 48 ± 6 hours | 48 ± 6 hours
  Determined by a dedicated core imaging laboratory, blinded to clinical data and timing of the CT studies. Scores range from 0-40 with 0 meaning no obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, MD, MS, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will consider requests of scientific merit

REFERENCES:
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Background] Hassan SM, Nardelli P, Minhas JK, Ash SY, Estepar RSJ, Antkowiak MC, Badlam JB, Piazza G, Estepar RSJ, Washko GR, Rahaghi FN. CT imaging determinants of persistent hypoxemia in acute intermediate-risk pulmonary embolism. J Thromb Thrombolysis. 2023 Jul;56(1):196-201. doi: 10.1007/s11239-023-02813-x. Epub 2023 May 4. PMID 37140805
- [Background] Klok FA, Piazza G, Sharp ASP, Ni Ainle F, Jaff MR, Chauhan N, Patel B, Barco S, Goldhaber SZ, Kucher N, Lang IM, Schmidtmann I, Sterling KM, Becker D, Martin N, Rosenfield K, Konstantinides SV. Ultrasound-facilitated, catheter-directed thrombolysis vs anticoagulation alone for acute intermediate-high-risk pulmonary embolism: Rationale and design of the HI-PEITHO study. Am Heart J. 2022 Sep;251:43-53. doi: 10.1016/j.ahj.2022.05.011. Epub 2022 May 16. PMID 35588898
- [Background] Piazza G. Advanced Management of Intermediate- and High-Risk Pulmonary Embolism: JACC Focus Seminar. J Am Coll Cardiol. 2020 Nov 3;76(18):2117-2127. doi: 10.1016/j.jacc.2020.05.028. PMID 33121720
- [Background] Rahaghi FN, San Jose Estepar R, Goldhaber SZ, Minhas JK, Nardelli P, Vegas Sanchez-Ferrero G, De La Bruere I, Hassan SM, Mason S, Ash SY, Come CE, Washko GR, Piazza G. Quantification and Significance of Pulmonary Vascular Volume in Predicting Response to Ultrasound-Facilitated, Catheter-Directed Fibrinolysis in Acute Pulmonary Embolism (SEATTLE-3D). Circ Cardiovasc Imaging. 2019 Dec;12(12):e009903. doi: 10.1161/CIRCIMAGING.119.009903. Epub 2019 Dec 17. No abstract available. PMID 31842589